CLINICAL TRIAL: NCT01117402
Title: Phase II Study Evaluating the Role of Tomotherapy- Based Intensity Modulated Radiotherapy and Brachytherapy in Postsurgery Recurrent Carcinoma Cervix
Brief Title: Tomotherapy in Postsurgery Recurrent Carcinoma Cervix
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Dr Reena Engineer, Tata Memorial Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 588
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Postsurgery Recurrent Carcinoma Cervix
Keywords: recurrent carcinoma cervix; Vault carcinoma; Tomotherapy; Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Radiotherapy — Patients will receive external radiation therapy using IMRT to pelvis. Treatment volume (CTV, vault and uninvolved pelvic nodes) will receive a dose of 50-56Gy over 25-28# and gross pelvic nodes will receive 55-62Gy over 25-28 fractions over 5 weeks. Pre RT daily MV CT imaging would be done on Tomotherapy to look and correct for any set up error or anatomic variations.
  Chemotherapy will be given weekly - cisplatin 40mg/m2 with prechemo medication. After completion of IMRT all patients will be evaluated for boost to vaginal vault with interstitial template brachytherapy to a dose of 16-20 Gy with HDR in 4-5 fractions. Patients not eligible for brachytherapy will get additional boost to vault and parametrium by EBRT to a dose of 15-20Gy in 6-8 fractions.
  Other Names: IMRT; Template brachytherapy

SUMMARY:
Radiotherapy is the most appropriate treatment for postoperative recurrent carcinoma cervix. However it is technically difficult to deliver adequate doses of RT due to presence of small intestines in the radiation area; thus disease control rates are poor and complication rates are high with conventional radiotherapy. Use of IMRT and brachytherapy for these cases allows for increasing dose to the tumor while sparing normal structures. It is expected that the use of a combination of IMRT & brachytherapy will achieve higher disease control rates and decrease the complication rates.

DETAILED DESCRIPTION:
SPECIFIC OBJECTIVES:

1. To evaluate the efficacy of combination of intensity-modulated radiotherapy (IMRT) and brachytherapy in delivering dose escalated radiotherapy in postoperative residual / recurrent cases of carcinoma cervix, in terms of local control proportion and progression free survival (PFS)
2. To study the late and acute toxicities associated with this treatment.
3. Dosimetric comparison of Tomotherapy and conventional IMRT

DESIGN: Prospective, phase II study.

STUDY POPULATION: All patients of age < 65 years diagnosed with postsurgery recurrent squamous cell carcinoma cervix without previous history of radiotherapy.

STUDY SIZE: 90 patients

METHODOLOGY: Ninety cases of cervical cancer with postsurgery recurrence limited to the pelvis will be screened and taken for study if eligible after taking the informed consent.

Patients will receive external radiation therapy using IMRT to pelvis with additional dose of localized radiotherapy boost with brachytherapy to the vault with weekly concurrent chemotherapy.

The local recurrence rate and 5 year disease free survival rate of all the patients will be studied.

PROJECT PERIOD:

Total project period : 5 years Recruitment, Data collection : 4 years Complete analysis of data : 1 year

STUDY SITE: Tata memorial centre

ELIGIBILITY:
Inclusion Criteria:

. Only histologically proven postoperative recurrence of squamous carcinoma of cervix following hysterectomy >3 months without adjuvant treatment

* Patients below 65 years of age and with KPS >70%.
* Patients with disease confined to the pelvis, based on CT/MRI/PET Scan
* Normal ECG and cardiovascular system
* Normal hematological parameters
* Normal renal and liver function tests

Exclusion Criteria:

* Previous chemotherapy or radiotherapy to the pelvis
* Pelvic LN >3cm in size
* Presence of disease outside the pelvis (Paraortic nodes, distant metastasis)
* Bilateral hydronephrosis
* Co-morbid conditions like uncontrolled Diabetes Mellitus or medical renal disease
* Medical or Psychological condition that would preclude treatment
* Patient unreliable for treatment and follow-up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the utility of intensity-modulated radiotherapy (IMRT) in delivering dose escalated radiotherapy in postoperative recurrent cases of carcinoma cervix, in terms of local control | 3 Years
  Progression free survival of all patients

SECONDARY OUTCOMES:
To study the late toxicities associated with this treatment | 3 Years
  Side effects of radiotherapy and chemotherapy will be recorded at baseline, during treatment, at 6 and 12 months and annually thereafter according to the RTOG scales

CONTACTS AND LOCATIONS:
Overall Officials: Reena Engineer, MD, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India